CLINICAL TRIAL: NCT02451007
Title: Evaluation of the Effect of Lurbinectedin (PM01183) on Cardiac Repolarization (QTc Duration) in Patients With Selected Solid Tumors
Brief Title: Evaluation of the Effect of Lurbinectedin (PM01183) on Cardiac Repolarization in Patients With Selected Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PM1183-B-005-14-QT
Record Dates: First submitted 2015-05-12; First posted 2015-05-21 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Solid Tumors
MeSH Terms: interventions — PM 01183

ARMS (1):
- A (lurbinectedin) (Experimental): lurbinectedin (PM01183) 4 mg vials of powder for concentrate for solution for infusion
  Interventions: Drug: lurbinectedin (PM01183)

INTERVENTIONS:
Drug: lurbinectedin (PM01183)

SUMMARY:
Study to assess the potential effects of lurbinectedin (PM01183) at a therapeutic dose on the duration of the QTc interval, measured by electrocardiograms (ECGs), to characterize the PM01183 plasma concentration/QTc relationship, and to explore related ECG parameters in patients with selected solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated informed consent
* Normal cardiac conduction and function (centrally read)
* Blood pressure between 90 and 150 mmHg systolic, inclusive, and not higher than 90 mmHg diastolic.
* Specific serum electrolyte levels

Exclusion Criteria:

* Age > 65 years
* Performance status = 2 [Eastern Cooperative Oncology Group (ECOG)]
* Heart rhythm disturbances
* Significant ischemic coronary disease, heart failure, myocardial infarction, or unstable angina within the last six months.
* Prior exposure to anthracyclines at a cumulative dose of doxorubicin (or equivalent) > 450 mg/m²

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Dana Farber Cancer lnstitute, Boston, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas
- Spain (11):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complejo Hospitalario de Especialidades Virgen de La Victoria, Málaga
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitari I Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was nested into a multicenter clinical trial with a competitive recruitment. From August 2015 to June 2016, a total of 39 evaluable patients at 12 sites in USA and Spain were included in this QT evaluation study with baseline and one or more postbaseline Electrocardiogram (ECG) assessments available.
Groups:
- Group A - Lurbinectedin (PM01183): lurbinectedin (PM01183) is presented as a lyophilized powder for concentrate for solution for infusion with strength of 4 mg / vial.
  Lurbinectedin was administered at a dose of 3.2 mg/m² given as a 1-hour i.v. every three weeks (q3wk) (three weeks = one treatment cycle). QTc interval duration was assessed when the patient was treated with lurbinectedin for the first time.
Period: Overall Study
Arm/Group | Group A - Lurbinectedin (PM01183)
Started | 39
Completed | 32
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Group A - Lurbinectedin (PM01183)
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 56 [28 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
  Spain | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in QTcF (QT Corrected According to Fridericia's Formula)
Description: ΔQTCF (Change in QTcF); EOI (end of infusion); LSM (Least Square Means); PK (Pharmacokinetic(s)).
  On Day 1 (D1) of Cycle 1 (C1), LSM ΔQTcF should have low difference values, without any clear trend to change with time.
  Therefore, the upper bound (UB) of the (two-sided) 90%Confidence Interval (CI) at all time points had to be less than the protocol-specified cut-off of 20 ms at each time point. If so, non-inferiority of any ECG time point to baseline with respect of QTc prolongation could be concluded
Time Frame: Scheduled post-baseline ECG time points were taken 5-10 min before their time-matched PK samples: i.e., 5 min before EOI, 30 min, 1, 3, 24, 72 and 168 hours after EOI of Cycle 1, and 5 min before EOI, 30 min, 1, 3 and 168 hours after EOI of Cycle 2.
Measure: Least Squares Mean (90% Confidence Interval); unit: ms (Milliseconds)
Arm/Group | Group A - Lurbinectedin (PM01183)
Number analyzed (Participants) | 39
ms (Milliseconds)
  Cycle 1 - 5 min before EOI | 3.32 [1.12 to 5.51]
  Cycle 1 - 30 min after EOI | 1.76 [-0.41 to 3.93]
  Cycle 1 - 1 hour after EOI | 1.84 [-1.02 to 4.69]
  Cycle 1 - 3 hour after EOI | 1.32 [-1.40 to 4.05]
  Cycle 1 - 24 hour after EOI | -8.24 [-11.2 to -5.26]
  Cycle 1 - 72 hour after EOI | -12.4 [-15.4 to -9.39]
  Cycle 1 - 168 hour after EOI | -5.20 [-7.98 to -2.41]
  Cycle 2 - Before start of infusion | -0.46 [-3.27 to 2.35]
  Cycle 2 - 5 min before EOI | 2.25 [-1.18 to 5.68]
  Cycle 2 - 30 min after EOI | 2.32 [-1.02 to 5.66]
  Cycle 2 - 1 hour after EOI | 2.73 [-1.08 to 6.54]
  Cycle 2 - 3 hour after EOI | 5.39 [1.17 to 9.60]
  Cycle 2 - 168 hour after EOI | -4.22 [-7.36 to -1.08]

2. Secondary Outcome: Relationship Between ΔQTcF and Time-matched Lurbinectedin Plasma Concentrations (Plasma Concentration)
Description: ΔQTcF (Change from Baseline in QT Corrected According to Fridericia's Formula); CI (Confidence Interval); Cmax (Maximum Plasma Concentration).
  Table below details the results of the linear mixed effects model to quantify the relationship between the lurbinectedin plasma concentrations and ΔQTcF and Predicted ΔQTcF and 90% CI at mean lurbinectedin Cmax.
Time Frame: Through study completion, each patient had to be followed for 2 cycles (1 cycle =3 weeks)
Measure: Mean (90% Confidence Interval); unit: Microgram/milliliter (μg/mL)
Arm/Group | Group A - Lurbinectedin (PM01183)
Number analyzed (Participants) | 39
Microgram/milliliter (μg/mL) | 2.06 [1.42 to 2.71]

3. Secondary Outcome: Relationship Between ΔQTcF and Time-matched Lurbinectedin Plasma Concentrations (Predicted ΔQTcF)
Description: as for outcome 2
Time Frame: Through study completion, each patient had to be followed for 2 cycles (1 cycle =3 weeks)
Measure: Mean (90% Confidence Interval); unit: Milliseconds (ms)
Arm/Group | Group A - Lurbinectedin (PM01183)
Number analyzed (Participants) | 39
Milliseconds (ms) | 2.94 [0.79 to 5.10]

4. Secondary Outcome: Relationship Between ΔQTcF and Time-matched Lurbinectedin Plasma Concentrations (Intercept)
Description: as for outcome 2
Time Frame: Through study completion, each patient had to be followed for 2 cycles (1 cycle =3 weeks)
Measure: Number (90% Confidence Interval); unit: Unitless
Arm/Group | Group A - Lurbinectedin (PM01183)
Number analyzed (Participants) | 39
Unitless | -6.40 [-8.44 to -4.35]

ADVERSE EVENTS:
Time Frame: Through study completion, each patient had to be followed for 2 cycles (1 cycle =3 weeks)
Groups:
- Group A - Lurbinectedin (PM01183): lurbinectedin (PM01183) is presented as a lyophilized powder for concentrate for solution for infusion with strength of 4 mg / vial.
  Lurbinectedin was administered at a dose of 3.2 mg/m² given as a 1-hour i.v. every three weeks (q3wk) (three weeks = one treatment cycle).
Arm/Group | Group A - Lurbinectedin (PM01183)
All-Cause Mortality (participants affected / at risk) | 13/39
Serious Adverse Events (participants affected / at risk) | 9/39
Other Adverse Events (participants affected / at risk) | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Lurbinectedin (PM01183) (N=39)
Blood calcium decreased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
General physical health deterioration (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Device related infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Lurbinectedin (PM01183) (N=39)
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 6
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Fatigue (General disorders) | 15
Pyrexia (General disorders) | 4
Insomnia (Psychiatric disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less